CLINICAL TRIAL: NCT01034683
Title: Phase 3 Study of Lobaplatin，5-Fluorouracil and Leucovorin for the Treatment of Recurrent or Metastatic Esophageal Carcinoma
Brief Title: Study of Lobaplatin，5-Fluorouracil and Leucovorin for the Treatment of Esophageal Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Taian Cancer Hospital (Other)
Responsible Party: Taian Cancer Hospital, Taian Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TACH2009001
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2010-01-05 (Estimated); Status verified 2009-12

CONDITIONS: Esophageal Carcinoma
MeSH Terms: conditions — Esophageal Neoplasms | interventions — lobaplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Esophageal Carcinoma (Experimental)
  Interventions: Drug: lobaplatin , 5-FU ,leucovorin

INTERVENTIONS:
Drug: lobaplatin , 5-FU ,leucovorin — Participants received 2-hour lobaplatin (30 mg/m2 on day 1) and a 2-hour infusion of leucovorin (LV; 200 mg/m2 on days 1-5) followed by a 4-hour infusion of 5-FU (650 mg/m2 on days 1-5). Treatment was repeated every 21 days.
  Other Names: LBP ,5-FU,LV

SUMMARY:
The purpose of this study is to evaluate the efficacy and the toxicity of lobaplatin, 5-fluorouracil (5-FU) and leucovorin in patients with esophageal carcinoma.

DETAILED DESCRIPTION:
patients with metastatic or recurrent esophageal cancer have a particularly poor prognosis .The overall 5-year survival rate for patients with newly diagnosed esophageal cancer is under 10%. Metastatic esophageal carcinoma is an incurable disease and due to the lack of effective therapies to manage this disease,the median survival is only 6 to 8 months Chemotherapy which is one of the most effective treatment so far is used as part of combined modality therapy for locally advanced diseases or as a palliative treatment for metastatic diseases.Lobaplatin is the third generation of platinum.Phase Ⅱclinical trials indicate that lobaplatin is effective for esophageal cancer, ovarian cancer, breast cancer and small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven squamous cell carcinoma of the esophagus(include cardiac cancer)
* Newly diagnosed patients should be unable or unwilling to surgery
* Recurrence after surgery must have no adjuvant chemotherapy or radiotherapy are allowed
* Patients are required to have dimensionally measurable disease,with an objective measurable focus:preferably the use of spiral computed tomography(CT)and measurements of maximum diameter≥1cm.
* Cooperative Oncology Group performance status 0-2 or KPS score ≥60,survival time ≥3 months
* Neutrophils(ANC)≥1.5×109/L; blood platelets counts(BPC)≥80×109/L
* Hemoglobin(Hgb)≥90g/L ,serum total bilirubin ≤1.0 times the upper normal limit(ULN): alanine aminotransferase and glutamic-oxalacetic transaminase (ALT and AST)≤2.5 ULN
* Serum creatinine (Cr)≤1.5ULN

Exclusion Criteria:

* pregnant or nursing women;
* Female patients at child-bearing age, without taking effective contraceptive methods;
* patients who have pathologic confirmation of other types of tumors (eg, leiomyosarcoma, malignant lymphoma) rather than esophageal cancer;
* patients with tumors other than esophageal cancer ,except cervical carcinoma in situ and skin basal cancer or squamous cell carcinoma received adequate treatment;
* patients with cerebral or meningeal metastasis, intestinal obstruction, or symptomatic pathologic changes of peripheral nerve,NCIC-CTG standard >grade 2
* patients with serious complications such as: serious heart disease remained unstable after treatment, or myocardial infarction, congestive heart failure, unstable angina, frank pericardial effusion or unstable arrhythmias in 6 months before being enrolled into the group; confirmed neuropathy or psychosis, including dementia or epilepsia; uncontrolled infection;active disseminated intravascular coagulation;uncontrolled diabetes, fasting serum glucose> 7.8mmol / L

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
objective response rate(ORR) time to progression (TTP) toxicities | 12/31/2010

SECONDARY OUTCOMES:
1-year survival rate KPS score | 12/31/2009

CONTACTS AND LOCATIONS:
Overall Officials: Lin Guan, Study Chair — Taian Cancer Hospital
Locations (1):
- Taian Cancer Hospital, Taian, Shandong, China